CLINICAL TRIAL: NCT06697314
Title: Prospective, Multicenter, Multi-national, Single Arm Trial Evaluating the Efficacy, Safety and Long Term Functional Outcomes of Percutaneous Mechanical Aspiration Thrombectomy for Treatment of Acute Pulmonary Embolism Using the AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Brief Title: Evaluating the Efficacy, Safety and Long Term Functional Outcomes of Percutaneous Mechanical Aspiration Thrombectomy for Treatment of Acute Pulmonary Embolism Using the AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System
Acronym: RECOVER-AV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-EVT-01
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Acute Pulmonary Embolism (PE); Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm Study - Use of AngioDynamics' AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 PE (Experimental): Prospective single-arm trial reporting the efficacy, safety, and long-term functional outcomes of percutaneous mechanical aspiration thrombectomy using the AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System for the treatment of acute pulmonary embolism.
  Interventions: Device: AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System

INTERVENTIONS:
Device: AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System — Single Arm Study - Use of AngioDynamics' AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 for the treatment of acute pulmonary embolism
  Other Names: thrombectomy; mechanial aspiration

SUMMARY:
To evaluate the efficacy, safety, and long-term functional outcomes of percutaneous mechanical aspiration thrombectomy using the AlphaVac Multipurpose Mechanical Aspiration (MMA) F1885 System for the treatment of acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, CTPA-proven acute PE with a maximum duration of symptoms of 14 days, showing a filling defect in at least one main or proximal lobar pulmonary artery
* RV/LV diameter ratio ≥ 1.0 assessed by CTPA
* Serum troponin levels above upper limit of normal as per hospital policy
* ≥ 18 years of age
* At least one of the following:

  1. Electrocardiogram (ECG)-documented tachycardia with heart rate ≥ 100 BPM, not due to hypovolemia, arrhythmia or sepsis
  2. Systolic blood pressure ≤ 110mmHg for at least 15 minutes
  3. Respiratory rate > 20 breaths per minuted. Oxygen saturation on pulse oximetry (SpO2) < 90% (or partial arterial oxygen pressure < 60 mmHg) at rest while breathing room air
  4. Known history of heart failure
* Willing and able to provide written informed consent prior to receiving study specific procedures.

Exclusion Criteria:

* A contraindication to therapeutic anticoagulation
* Any comorbid diagnosis consistent with a life expectancy of less than 1 year (e.g., stage 4 cancer)
* Known serious, uncontrolled sensitivity to radiographic agents
* Cardiac arrest within last 14 days without documented evidence of recovery of conscious level to Glasgow Coma Scale >12
* Indication for ECMO
* Pregnant or breastfeeding
* Participation in another investigational drug or device study that study may confound the results of this study. Studies requiring extended follow-up for products that were investigational but have since become commercially available are not considered investigational studies.
* Other medical, social, or psychological conditions that, in the opinion of the Investigator, precludes the patient from appropriate consent, could limit the patient's ability to participate in the study, including compliance with follow- up requirements, or that could impact the scientific integrity of the study.
* History of congenital or acquired bleeding disorder predisposing to hemorrhagic state
* Platelet count < 100,000/μL
* Any advanced reperfusion therapy for pulmonary embolism within 30 days of the index procedure (e.g lysis, surgery, catheter intervention)
* A known clot in transit
* IVC filter
* A do not resuscitate limitation at inclusion in the study
* Deprived of liberty or under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in RV/LV ratio | 48 hours
  Reduction in RV/LV ratio between baseline and 48 hours post-procedure assessed by paired computed tomography pulmonary angiography (CTPA)
Incidence of Adverse Events [Safety and Tolerability] | 12 months
  The primary safety endpoint is the incidence of adverse events by type and seriousness through 12 months. The number and proportion of subjects who experienced at least one adverse event will be summarized, and the 95% confidence interval of the proportion will be presented.

SECONDARY OUTCOMES:
Reduction in clot burden | 48 hours
  • Reduction in clot burden (measured by refined Modified Miller Index score) between baseline and 48 hours post-procedure assessed by paired CTPA
Use of thrombolytics | 48 hours
  Use of thrombolytics within 48 hours of the index procedure
Change in Biomarkers | 48 hours
  Change in troponin, BNP, and D-dimer from baseline to 48 hours post-procedure
Composite Major Adverse Events | 7 days
  * Composite Major Adverse Events within 7 days of the index procedure
    1) PE-related death/deterioration:
  * Death
  * Cardiac Arrest
  * Institution of new vasopressors
  * ECMO
  * Mechanical ventilation
    2) Device-related death/deterioration:
  * Death
  * BARC 3a/3b/3c/-5 Major Bleeding
  * Clinical Deterioration
  * Pulmonary Vascular Injury
  * Peripheral Vascular Injury
  * Cardiac Injury
  * Stroke
Individual Major Adverse Events | 7 days
  Individual Major Adverse Events within 7 days of the index procedure
  * PE-related Death
  * PE-related Cardiac Arrest
  * PE-related institution of new vasopressors
  * PE-related ECMO
  * mechanical ventilation
  * device-related Death
  * device-related Major Bleeding
  * device-related Clinical Deterioration
  * device-related Pulmonary Vascular Injury
  * device-related Peripheral Vascular Injury
  * device-related Cardiac Injury
  * device-related Stroke
Days in ITU | 7 days
  Days in ITU post-index procedure admission
All-cause mortality | 30 days
  All-cause mortality within 30 days of the index procedure
PE-related mortality | 30 days
  • PE-related mortality within 30 days of the index procedure
Device-related Serious Adverse Events | 30 days
  Device-related Serious Adverse Events (SAEs) within 30 days of the index procedure
Days In-patient | 30 days
  Number of days in-patient on index procedure admission
Hospital readmission | 30 days
  Hospital readmission rate through 30 days
Symptom burden exercise test | 30 days
  6 minute walking test (MWT) at 30 days post-procedure
Symptom burden classification | 30 Days
  New York Heart Association (NYHA) classification at 30 Days post-procedure
Functional outcome review | 30 Days
  PROMs at 30 Days post-procedure:
  * PROMIS Scale v1.2 - Global Health
    - PEmb-QoL
  * Post-VTE Functional Status Scale
  * PROMIS Short Form v2.0 - Pain Intensity 3a
  * PROMIS Short Form v1.0 - Dyspnea Severity 10a
  * PHQ-9
  * GAD-7
Symptomatic PE recurrence | 30 days
  Symptomatic PE recurrence at 30 days post-procedure
Symptom burden exercise test | 6 months
  6 minute walking test (MWT) at 6 months post-procedure
Symptom burden classification | 6 months
  New York Heart Association (NYHA) classification at 6 months post-procedure
PE-related readmission | 12 months
  - PE-related hospital readmission rate through 12 months post-procedure
Symptom burden exercise test | 12 months
  6 minute walking test (MWT) at 12months post-procedure
Symptom burden classification | 12 months
  New York Heart Association (NYHA) classification at 12 months post-procedure
Functional outcome review | 12 months
  PROMs at 12 months post-procedure:
  * PROMIS Scale v1.2 - Global Health
    - PEmb-QoL
  * Post-VTE Functional Status Scale
  * PROMIS Short Form v2.0 - Pain Intensity 3a
  * PROMIS Short Form v1.0 - Dyspnea Severity 10a
  * PHQ-9
  * GAD-7
CTEPH Diagnosis | 12 months
  Diagnosis of chronic thromboembolic pulmonary hypertension (CTEPH) at 12 months post-procedure

OTHER OUTCOMES:
Cardiac MRI | 12 months
  • Cardiac MRI at 12-months post-procedure (for up to 100 patients) to assess:
  * RA/RV dimension and function
  * Signs of RV fibrosis
  * Pulmonary parenchymal function and abnormalities
  * Pulmonary vascular structure
  * Tricuspid regurgitation severity
  * Ventricular Septal motion characteristics
Peak Oxygen Consumption | 12 months
  • Peak Oxygen consumption (for up to 100 patients): PVO2 measured during cardiopulmonary exercise test at 12 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sharp, Principal Investigator — University College Dublin, Rep. of Ireland; Erik Klok, Principal Investigator — Leiden UMC, The Netherlands
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.angiodynamics.com/studies/recover-av/